CLINICAL TRIAL: NCT00934869
Title: Swelling or Malrotation of Metacarpal Shaft Fractures in the Evaluation of Rotational Deformity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: LUR01-CTIL -HMO
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Metacarpal Shaft Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metacarpal Shaft Fractures

SUMMARY:
Rotational deformity or malunion causes the most significant functional deficit in these common fractures. The evaluation of the rotation may be performed with the metacarpophalangeal joints flexed although postoperative swelling may not enable this examination with flexion of the fingers. Furthermore, it has been shown that swelling may cause rotation of the digit itself. The investigators propose that the swelling may cause a mistake in the estimation of rotation, during surgery and early follow up period. This is of special importance when open reduction and rigid fixation is performed.

Methods:

Prospective analysis of XX isolated metacarpal fractures treated, in YY patients was performed. End-on view of the finger-nail was taken with a digital camera on the day of OR, at 2 weeks and at 1 year. The photos were taken on a standard apparatus and from a distance of XX cm and evaluated using ZZ software in comparison with photos taken of the other hand, according to the involved digit. Range of motion, type of fracture and type of fixation were compared.

ELIGIBILITY:
Inclusion Criteria:

1. isolated metacarpal fractures in one hand- fingers 2, 3, 4, 5
2. treated with cast or surgical treatment , closed or open reduction

Exclusion Criteria:

1. multiple fractures simultaneously
2. fractures in both hands
3. former fracture in one of the fingers, two palms,metacarpal,proximal phalanx (with exception of the thumb)
4. open fracture, open wounds, infection
5. pregnancy, inability performing full x-ray follow up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and Women with isolated metacarpal fractures
Sampling Method: Non-Probability Sample
Dates: Start 2009-08; Primary Completion 2015-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel